CLINICAL TRIAL: NCT02310009
Title: IL-1RA, Acute Exercise, and Beta-cell Function
Acronym: ANEX
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI relocated to a different country and coI moved to a different lab.
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Solomon, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ANEX
Record Dates: First submitted 2014-12-02; First posted 2014-12-05 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Exercise; IL-1RA; Beta-cell function; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity | interventions — Interleukin 1 Receptor Antagonist Protein; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (CON) (Experimental): Placebo will be administered as a subcutaneous injectable bolus, the day prior to the repeated measurement of beta-cell function.
  Interventions: Behavioral: Control (CON)
- Anakinra (AN) (Experimental): 100 mg of Kineret (Anakinra) will be administered as a subcutaneous injectable bolus, the day prior to the repeated measurement of beta-cell function.
  Interventions: Drug: Anakinra (AN)
- Exercise (EX) (Experimental): 1 hour of cycling exercise will be performed at 75% VO2max, the day prior to the repeated measurement of beta-cell function.
  Interventions: Behavioral: Exercise (EX)
- Anakinra + Exercise (ANEX) (Experimental): 100 mg of Kineret (Anakinra) will be administered as a subcutaneous injectable bolus followed by 1 hour of cycling exercise at 75% VO2max, the day prior to the repeated measurement of beta-cell function.
  Interventions: Drug: Anakinra (AN); Behavioral: Exercise (EX)

INTERVENTIONS:
Drug: Anakinra (AN)
  Arms: Anakinra (AN); Anakinra + Exercise (ANEX)
Behavioral: Exercise (EX)
  Arms: Anakinra + Exercise (ANEX); Exercise (EX)
Behavioral: Control (CON)
  Arms: Control (CON)

SUMMARY:
Subjects (N=48) with poorly-controlled type 2 diabetes (HbA1c>7%) will be assigned to one of the 4 following interventions in a randomised, parallel group design: [I] Control (placebo injection; no exercise), [II] Anakinra (100 mg subcutaneous injection of human recombinant interleukin-1 receptor antagonist), [III] Exercise (1 h cycle ergometry at 75% VO2max), [IV] Anakinra + Exercise. Pancreatic beta-cell function (plasma insulin responses) will be measured before and after each intervention using a hyperglycemic clamp (5.4 mM above basal glucose) combined with GLP-1 infusion (0.5 pmol/kg/min) and arginine injection (5 g bolus).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with HbA1c >7%

Exclusion Criteria:

* HbA1c >7%
* Age <30 or >80 y
* BMI <25 or >40 kg/m2
* Pregnancy
* Evidence of chronic haematological/renal/hepatic/pulmonary/heart disease
* >2kg weight change in prior 6 months
* Alcohol consumption (men: >14 drinks/week; women: >7 drinks/week)
* Smoking
* Physical activity of >150 min/week
* Contraindication to exercise
* Contraindication to use of anakinra

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Estimated); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Beta-cell function | 1 day after intervention
  A hyperglycemic clamp will be performed combined with glucagon-like peptide(GLP)-1 infusion and arginine injection. The primary outcome is the insulin secretory response to glucose, GLP-1, and arginine.

SECONDARY OUTCOMES:
Glucose disposition | 1 day after intervention
  The glucose disposal rate during hyperglycemic clamp

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Solomon, PhD, Principal Investigator — Rigshospitalet & University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark